CLINICAL TRIAL: NCT03626753
Title: Comparison of Two Routes of Administration of a Multimodal Analgesic Protocol in Postoperative Cesarean Section Oral vs Intravenous
Brief Title: Comparison of Two Routes of Administration of a Multimodal Analgesic Protocol in Postoperative Cesarean Section
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Centre de Maternité de Monastir (Other)
Responsible Party: Principal Investigator, Fethi Jebali, Medical doctor, clinical professor of Anesthesiology and intensive care medecine, Centre de Maternité de Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMNMonastir
Record Dates: First submitted 2018-07-31; First posted 2018-08-13 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Cesarean Section; Complications, Wound, Infection (Following Delivery); Postoperative Pain; Spinal Anaesthesia During the Puerperium
Keywords: Pain; multimodal; analgesia; postoperative; cesarean section; obstetric; Agents; Physiological effects of drugs; opioid; Paracetamol; NSAIDs
MeSH Terms: conditions — Wounds and Injuries; Infections; Pain, Postoperative; Pain; Agnosia | interventions — Nefopam; Acetaminophen; Tablets; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Group (Active Comparator): received in post operative period oral analgesia ( "nefopam (Acupan)" 20mg/6h, "piroxicam (piroxan)" 40mg/24h," Acetaminophen (paracetamol)" 1g/6h)
  Interventions: Drug: Nefopam 20 MG/ML; Drug: "Acetaminophen, (paracetamol)" 500Mg Tab; Drug: (Piroxicam "piroxan") 20 MG Oral Tablet
- Intravenous group (Active Comparator): received in post operative period intravenous analgesia ( "nefopam (Acupan)" 20mg/6h, "piroxicam (piroxan)" 40mg/24h," Acetaminophen (paracetamol)" 1g/6h)
  Interventions: Drug: "Nefopam (Acupan)" 20 MG/ML Injectable Solution; Drug: (Acetaminophen "paracetamol") IV Soln 10 MG/ML; Drug: (Piroxicam "piroxan") 20Mg/1mL Injection

INTERVENTIONS:
Drug: Nefopam 20 MG/ML — given by Oral route the dose of 20mg every 6 hours.
  Other Names: 2 ampoule
  Arms: Oral Group
Drug: "Nefopam (Acupan)" 20 MG/ML Injectable Solution — given by intravenous route at the dose of 20mg every 6 hours.
  Other Names: 2 ampoule
  Arms: Intravenous group
Drug: "Acetaminophen, (paracetamol)" 500Mg Tab — 2 tablets of "Acetaminophen (paracetamol)" 500Mg Tab administrated orally every 6 hours.
  Other Names: 2 tablets
  Arms: Oral Group
Drug: (Acetaminophen "paracetamol") IV Soln 10 MG/ML — Acetaminophen IV Soln 10 MG/ML, 1g paracetamol administrated intravenously every 6 hours.
  Other Names: 1 ampoule: 1g
  Arms: Intravenous group
Drug: (Piroxicam "piroxan") 20 MG Oral Tablet — 2 tablets of "piroxicam (piroxan)" administrated orally once per 24 hours.
  Other Names: 2 tablets
  Arms: Oral Group
Drug: (Piroxicam "piroxan") 20Mg/1mL Injection — 2 ampoules of (piroxicam "piroxan") administrated intravenously once per 24 hours.
  Other Names: 2 ampoules
  Arms: Intravenous group

SUMMARY:
Many drugs with various mechanisms of action are used for postcaesarean pain relief. Although the response to pain relief is sometimes believed to be individual, it is very important to establish the most effective with the least adverse effects type of oral analgesia for women after caesarean section. Optimal pain control post-caesarean section will benefit not only the mother and her baby, but also a healthcare system. Optimal pain control may shorten the time spent in hospital after caesarean section and, therefore, reduce healthcare costs.

DETAILED DESCRIPTION:
Pain after cesarean section (CS), usually described as strong, is an obstacle to good mother-child interaction and post-operative rehabilitation. Its management is important for a quick recovery and allow the mother to take care and link with her newborn. Currently, intrathecal opioids are the most commonly used technique and provide the foundation for post-cesarean analgesia. This technique combined with multimodal analgesia reduces the doses of morphine consumed, including these side effects. Spinal anesthesia is the standard anesthetic technique for caesarean section; it offers several advantages including the possibility of prescribing oral analgesics. An ideal analgesic protocol is one that is simple to implement, cost-effective, and has minimal impact on the work staff. It would have a good safety profile, a low incidence of side effects and complications, and respond to wide inter-patient variability. It relieves the mother of high quality pain while having minimal interference with her, newborn care and anesthesia while allowing safe breastfeeding.

The aim of this work is to compare the quality of an multimodal oral analgesia with intravenous analgesia and to demonstrate non-inferiority of the oral route pain relieve in postoperative caesarean section period. The secondary objectives was to evaluate the maternal tolerance of the drugs (piroxicam, nefopam, paracetamol) used postoperatively of a caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant in singleton pregnancy with gestational age > 34 weeks
* American society of anesthesiologists (ASA) physical status I-II.

Exclusion Criteria:

* history of gastrointestinal disorders predisposing to bleeding disorders such as ulcerative colitis,
* Crohn's disease,
* gastrointestinal cancers or diverticulitis,
* an active peptic ulcer,
* an inflammatory gastrointestinal disorder or a gastrointestinal haemorrhage,
* parturients who present preeclampsia,
* premature delivery (<32 weeks),
* constitutional or acquired coagulopathy,
* An antecedent of hemorrhage of the delivery,
* a hemorrhagic complication postoperatively,
* Anemia (hemoglobin less than 8g / 100ml),
* conversion of spinal anesthesia into general anesthesia,
* women with severe medical conditions: renal failure (preoperative creatinine clearance <30ml / min), heart or liver failure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) pain | 24 hours postoperative
  from 0 - 10 (with 0 being no pain and 10 being the most severe pain imaginable) at rest and coughing or mobilization

SECONDARY OUTCOMES:
morphine consumption | 24 hours postoperative
  morphine consumption
sides effects | 24 hours postoperative
  the occurrence of any undesirable effects related to the administration of any of the 3 drugs (nausea, vomiting, diarrhea, malaise, hypotension, sweating, convulsion, dryness of the mouth, tachycardia, palpitations, vertigo, allergic reactions)
postoperative complications | 24 hours post operative
  The occurrence of a postoperative complication (postpartum haemorrhage, blood transfusion, hysterectomy, etc).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Maternité de Monastir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mahajan L, Mittal V, Gupta R, Chhabra H, Vidhan J, Kaur A. Study to Compare the Effect of Oral, Rectal, and Intravenous Infusion of Paracetamol for Postoperative Analgesia in Women Undergoing Cesarean Section Under Spinal Anesthesia. Anesth Essays Res. 2017 Jul-Sep;11(3):594-598. doi: 10.4103/0259-1162.206872. PMID 28928554
- [Background] Mkontwana N, Novikova N. Oral analgesia for relieving post-caesarean pain. Cochrane Database Syst Rev. 2015 Mar 29;2015(3):CD010450. doi: 10.1002/14651858.CD010450.pub2. PMID 25821010